CLINICAL TRIAL: NCT01913054
Title: Combined Use of Etomidate and Propofol in Painless Gastroscopy, a Multiple Center, Double Blinded, Randomized,Controled Study.
Brief Title: Combined Use of Etomidate and Propofol in Painless Gastroscopy.
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Jiangsu Nhwa Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: 2013072201
Record Dates: First submitted 2013-07-25; First posted 2013-07-31 (Estimated); Last update posted 2013-12-16 (Estimated); Status verified 2013-07

CONDITIONS: Safety of Gastroscopy
Keywords: Etomidate; Propofol; Painless gastroscopy
MeSH Terms: interventions — Fentanyl; Propofol

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Fentanyl & Propofol (Active Comparator): 0.02 ml/kg(1 μg/kg) fentanyl is diluted to 10 ml with normal saline and infused within 1 min, 4 min advance. 0.5 mg/kg(0.025 ml/kg) propofol is infused within 15 to 20 s. And then, depending on the randomized result, 0.5 mg/kg is given every time until the patient falls asleep. During the operation, 0.5 mg/kg is given when it is needed.
  Interventions: Drug: Fentanyl Injection; Drug: Propofol Injection
- fentanyl, propofol & etomidate (Experimental): 0.02 ml/kg(1 μg/kg) fentanyl is diluted to 10 ml with normal saline and infused within 1 min, 4 min advance. 0.5 mg/kg(0.025 ml/kg) propofol is infused within 15 to 20 s. And then, depending on the randomized result, 0.5 mg/kg etomidate is given every time until the patient falls asleep. During the operation, 0.5 mg/kg etomidate is given when it is needed.
  Interventions: Drug: Fentanyl Injection; Drug: Etomidate Fat Emulsion Injection; Drug: Propofol Injection

INTERVENTIONS:
Drug: Fentanyl Injection
Drug: Etomidate Fat Emulsion Injection
  Other Names: Fuerli
  Arms: fentanyl, propofol & etomidate
Drug: Propofol Injection
  Other Names: Jing'an

SUMMARY:
Gastroscopy, as a conventional examination for gastrointestinal tract disease, plays a very important role especially in early diagnosis and differential diagnosis of esophageal and gastric carcinoma. However, conventional gastroscopy is associated with several adverse effects (including throat discomfort, breath-holding, nausea, vomiting, laryngeal spasm and increased heart rate) due to which some patients are intolerant to this examination or even refuse the procedure due to fear of these effects. Recently, painless gastroscopy has been applied increasingly widely in outpatients to meet the increasing needs for comfortable medical care.

Painless gastroscopy is commonly performed under general anesthesia without establishing an artificial airway. This is associated with an even higher anesthetic risk than general anesthesia in the operating room due to more basic patient monitoring and life-supporting equipment, only one anesthetist to perform anesthesia, fatigue in anesthesia, the requirement for a high turnover rate, as well as limited understanding of a patient's condition. Therefore, the availability of sedatives and analgesics which can provide rapid onset, sufficient sedation and analgesia, a short recovery time and less adverse effects are the premise of performing painless gastroscopy. Currently, combined intravenous anesthesia with fentanyl and propofol, commonly used in the clinic, is still associated with a long duration of action, hypotension in some patients and prolonged recovery. Etomidate has been increasingly utilized for in-clinic diagnosis and treatment for procedures such as painless coloscopy and early induced abortion due to its rapid onset, rapid metabolism and minimal impact on the circulatory and respiratory systems. However, no study on combined intravenous anesthesia with fentanyl and etomidate for painless gastroscopy had previously been reported. The main purpose of this study is to explore the efficacy and safety of combined intravenous anesthesia with fentanyl and etomidate for painless gastroscopy compared with the combination of fentanyl and propofol in middle aged and elderly patients, and to provide reliable evidence for the implementation and promotion of comfortable medical care.

DETAILED DESCRIPTION:
There are 6 centers for this trial: General Hospital of Chinese People's Liberation Army, Chaoyang Hospital Attached to the Capital Medical University, The Second Affiliated Hospital of Harbin Medical University, Renmin Hospital of Wuhan University Hubei General Hospital, The Affiliated Hospital of Xuzhou Medical College, Hospital of Chinese Air Force.

ELIGIBILITY:
Inclusion Criteria:

* Preparing to take gastroscopy;
* Age:between 45 to 75 years old (middle-aged group: 45~59 years old; elderly group: 60~75 years old; the percentage of middle-aged group and elderly group are 60% and 40%, respectively);
* BMI: between 18 to 25 kg/m2;
* ASA classification: grade Ⅰ~Ⅱ.

Exclusion Criteria:

* Blood pressure before operation: >180 mm Hg or <90 mm Hg;
* ECG before operation: <50 beats per min;
* HGB before operation: <90 g/L;
* Infected with respiratory inflammation and not cured within 2 weeks;
* Sever heart, brain, pulmonary, heptic, renal diseases or diabetes;
* History of difficult airway or abnormal recovery from anesthesia before or difficult airway is predicted to occur ;
* Obvious electrolyte disturbance such as hyperkalemia;
* Treated with immunosuppressants such as hormones for a long time or prior inhibition of the adrenal cortex;
* Allergic to emulsion or opioids;
* Concomitant other sedatives or analgesics (including injectable or oral administration of treatment related to Chinese Traditional Patent Medicines);
* Suspected abuse of narcotic analgesics or sedatives;
* Patients for whom it is difficult to cooperate or communicate because of abnormalities of neuromuscular system or mental disorder.

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2450 (Estimated)
Dates: Start 2013-08; Primary Completion 2013-12 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
Blood pressure | baseline to 10 min after the operation, an expected average of 20 minutes
  Changes of blood pressure in each group will be recorded.

SECONDARY OUTCOMES:
Heart rate | baseline to the end of the operation, an expected average of 30 minutes
  Changes of heart rate in each group will be recorded.
Pulse Oxygen Saturation | baseline to the end of the operation, an expected average of 10 minutes
  Changes of pulse oxygen saturation in each group will be recorded.
Respiratory rate | baseline to the end of the operation, an expected average of 10 minutes
  Changes of respiratory rate in each group will be recorded

OTHER OUTCOMES:
efficacy of anesthesia | From the time when propofol is given to discharge, an expected average of 30 minutes
  The time when propofol is given is defined as the time when infusion of propofol is beginning.
  The time of discharge is defined as the time when Steward score of the patient ≥4.
Satisfaction | 10 minutes after the operation
  Record the satisfaction from the operator, the anesthetist and the patients
Recovery of anesthesia | 10 min, 15 min and 15 min after the operation
  Steward score was used to evaluate the recovery of anesthesia.
Recovery of orientation | 10 min, 15 min and 20 min after the operation
  MMSE scale is used to evaluate the recovery of orientation for each patient.
Comfort degree | 10 minutes after the operation
Adverse events | during the operation, an expected average of 10 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Weidong Mi, Senior, Principal Investigator — General Hospital of Chinese People's Liberation Army
Locations (6):
- China (6):
  - Chaoyang Hospital Attached to the Capital Medical University, Beijing, Beijing Municipality
  - General Hospital of Chinese Air Force, Beijing, Beijing Municipality
  - General Hospital of Chinese People's Liberation Army, Beijing, Beijing Municipality
  - The Second Affiliated Hospital of Harbin Medical University, Harbin, Heilongjiang
  - Renmin Hospital of Wuhan University Hubei General Hospital, Wuhan, Hubei
  - The Affiliated Hospital of Xuzhou Medical College, Xuzhou, Jiangsu